CLINICAL TRIAL: NCT03130725
Title: Comparison of Six Months Retention of Bonded Amalgam Sealants Versus Resin-based Sealants: A Randomized Controlled Trial
Brief Title: Retention of Bonded Amalgam Sealants Versus Resin-based Sealants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Farhan Raza Khan, Assistant Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 4445-CHS-ERC-16
Record Dates: First submitted 2017-04-22; First posted 2017-04-26 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Incipient Enamel Caries; Fissure, Dental
MeSH Terms: conditions — Dental Fissures

STUDY DESIGN:
Intervention Model Description: The study design will be parallel group, equivalence randomized controlled trial. Aim is to determine the equality of the Amalgam sealants retention compared to resin based sealants retention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amalgam sealant (Experimental): Amalgam sealant placed on incipient enamel caries and deep enamel fissures.
  Interventions: Procedure: Amalgam sealant
- Resin based sealant (Active Comparator): Resin based sealant placed on incipient enamel caries and deep enamel fissures.
  Interventions: Procedure: Resin based sealant

INTERVENTIONS:
Procedure: Amalgam sealant — Amalgam sealant placed on incipient enamel caries and deep enamel fissures.
  Arms: Amalgam sealant
Procedure: Resin based sealant — Resin based sealant placed on incipient enamel caries and deep enamel fissures.
  Arms: Resin based sealant

SUMMARY:
Dental caries, is one of the major public health problem in Pakistan. Dental sealants are known cost effective preventive measure of dental caries as compared to other preventive measures. Resin based sealants, is a proven treatment of pits and fissure sealants but retention is still problem. This trial will assess the use of amalgam sealants as an effective and retentive preventive measure in preventing dental caries in children as compared to the standard resin-based sealants. The findings of this randomized controlled trial will be used to raise awareness among the health care professionals, help them to choose amalgam sealants as an effective caries prevention method thereby reducing the burden of cost as amalgam is cheaper material compared to resin-based sealants.

The research question Is there any difference in the six months retention of bonded amalgam sealants compared to resin-based sealants among 12 to 16 years old children in Karachi

DETAILED DESCRIPTION:
Objective:

To compare the six month retention of bonded amalgam sealants with that of resin-based sealants among 12 to 16 year old children in Karachi

Methods:

The study design will be parallel group, equivalence randomized controlled trial. Aim is to determine the equality of the Amalgam sealants retention compared to resin based sealants retention.

Outcome:

The primary outcome will be Retention, divided into Complete Retention, Partial Retention and Dislodgement of the sealant material.

ELIGIBILITY:
Inclusion Criteria:

* Children of aged 12 to 16 years (male and female) who will visit to the study site and fulfilled the eligibility criteria
* Teeth should be caries free at the time of sealants placement. As Dental sealant is a preventive treatment it is placed in a caries free surface. Incipient carious lesions will also be included.
* Teeth should be completely erupted, as incomplete eruption of teeth is highly correlates to the partial retention of sealants.
* Children who will give assent to participate in a study and their parents will give consent.

Exclusion Criteria:

* Special needs children (because they need special attention of parents)
* Children who have blood disorder like (leukemia, lymphoma, and thalassemia)
* Persons with impaired vision, speech and hearing (because either they may not be able to respond to questionnaire or conducting baseline dental training will be difficult).

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-10-01 (Actual)

PRIMARY OUTCOMES:
Retention of sealant | Six months
  1. Complete retention, if the all the occlusal fissures were covered by the sealant.
  2. Partial retention, if some of occlusal fissures of a tooth showed loss of sealant.
  3. Complete failure, if sealant was missing from all the occlusal fissure of the tooth.

CONTACTS AND LOCATIONS:
Overall Officials: Samreen L Khowaja, MSc, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khan FR, Liaquat S, Rafique G, Azam SI, Hasan A. Bonded amalgam as a fissure sealant in low-income setting: A randomised controlled trial. J Pak Med Assoc. 2022 Feb;72(Suppl 1)(2):S3-S9. doi: 10.47391/JPMA.AKU-02. PMID 35202361